CLINICAL TRIAL: NCT05890209
Title: Optimizing Weight Loss. Can Continuous Glucose Monitoring Play a Role
Acronym: OWL-CGM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Nurul Zafirah Binti Mohd Hatta, Principal Investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200220068
Record Dates: First submitted 2023-04-28; First posted 2023-06-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Weight Loss; Obesity
MeSH Terms: conditions — Weight Loss; Obesity | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Weight Management group (PWM) (No Intervention): The group will receive a personalized diet and physical activity plan and five one-to-one online support meetings with a trained dietitian over the first 12 weeks of the program (in weeks 1, 2, 4, 8, and 12). The participants also will be given an evidence-based weight loss maintenance information booklet and advice (e.g.: dietary advice, physical activity recommendation, the importance of self-monitoring weight, diet, and physical activity). Participants will be asked to self-manage during weeks 12 - 24 and asked to maintain the diet, PA recommendations, and monitoring based on the advice and training provided in the first 12 weeks of the program.
- PWM + Continuous Glucose Monitoring (CGM) (Experimental): This group will receive the same support as the PWM group. The participants also will be given an evidence-based weight loss maintenance information booklet and advice (e.g.: dietary advice, physical activity recommendation, the importance of self-monitoring weight, diet, physical activity, and glucose level). In addition, participants will be provided with a CGM device and guidance on how to use this to support weight loss maintenance. They will be provided with CGM devices for the whole study duration.
  Interventions: Device: Continuous Glucose Monitoring device

INTERVENTIONS:
Device: Continuous Glucose Monitoring device — A small wearable transdermal sensor that tracks glucose levels in interstitial fluid by taking measurements at regular and frequent intervals throughout the day and night.
  Arms: PWM + Continuous Glucose Monitoring (CGM)

SUMMARY:
The goal of this clinical trial is to determine the potential effectiveness of adding Continuous Glucose Monitoring to a personalized weight loss maintenance program in improving weight loss maintenance.

The main questions it aims to answer are:

* What is the feasibility and acceptability of wearing a continuous glucose monitoring device in people maintaining weight loss?
* Is using continuous glucose monitoring will help to change the food and physical activity behavior in people maintaining weight loss?

Participants will be randomized into control and intervention groups where the researchers will compare the effects of wearing continuous glucose monitoring devices on behavior change in both groups.

DETAILED DESCRIPTION:
The study is a 24-week study conducted at the University of Glasgow. It is a randomized, non-blinded, feasibility trial with 48 adults randomized into one of two groups (24 adults in each group):

* Personalized Weight Management Group (PWM): The group will receive a personalized diet and physical activity plan and five one-to-one online support meetings with a trained dietitian over the first 12 weeks of the program (in weeks 1, 2, 4, 8, and 12). The participants also will be given an evidence-based weight loss maintenance information booklet and advice (e.g.: dietary advice, physical activity recommendation, the importance of self-monitoring weight, diet, and physical activity). Participants will be asked to self-manage during weeks 12 - 24 and asked to maintain the diet, PA recommendations, and monitoring based on the advice and training provided in the first 12 weeks of the program.
* PWM + CGM: This group will receive the same support as the PWM group. The participants also will be given an evidence-based weight loss maintenance information booklet and advice (e.g.: dietary advice, physical activity recommendation, the importance of self-monitoring weight, diet, physical activity, and glucose level). In addition, participants will be provided with a CGM device and guidance on how to use this to support weight loss maintenance. They will be provided with CGM devices for the whole study duration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Intentionally lost ≥5 kg within the past 6 months
* Have a BMI of >25kg/m2 prior to weight loss
* Have access to and be able to use a smartphone or tablet running iOS or Android and be able to use the Freestyle Libre app and MyFood24 app OR access and ability to use a telephone.
* Participants should be willing to use CGM.
* Participants must be able to read, understand and communicate in English

Exclusion Criteria:

* Have been diagnosed with Type 1 and Type 2 Diabetes
* Pregnant or planning pregnancy in the next 6 months, or currently breastfeeding.
* Participants who are currently on any pharmacological treatments for weight loss or any drugs may affect body weight.
* Participants who have previously had bariatric surgery for weight loss including gastric bypass and sleeve gastrectomy.
* Participants with known hypersensitivity to CGM sensors.
* Participants with any other serious medical condition, in the opinion of the investigators, would compromise their safety or adherence to the study.
* Participants diagnosed with an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or purging disorder).
* Participants who lack capacity or are unable to read or understand written or verbal instructions in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Research recruitment rate | 24 weeks
  The number of adults being recruited over the course of recruitment phase.
Research retention rate | 24 weeks
  Retention is the number of participants that remain till the end of the trial at the end of 24 weeks.
Adherence of CGM use | 24 weeks
  The proportion of days for which valid CGM data are obtained from the CGM group.
Changes in dietary intake | 24 weeks
  Dietary Intake monitored for 3 days at 0, 12, 24 weeks using the MyFood24 online diaries where the participants will have to log their daily dietary intake.
Changes in physical activity | 24 weeks
  Physical Activity level monitored objectively for a day using an accelerometer at 0, 12, 24 weeks.
Changes in weight | 24 weeks
  Weight will be monitored using weight scale from baseline Week 0, Week 12 and Week 24
Changes in body composition | 24 weeks
  Body composition will be measured using bioelectrical impedance at Week 0, 12, 24

SECONDARY OUTCOMES:
Qualitative evaluation of participant's experiences | 24 weeks
  Qualitative evaluation of participant's experiences will be conducted through a semi structured interview with 8-12 of participants
Changes in biomarkers of cardio-metabolic disease risk | 24 weeks
  Biomarkers measurement will be measured at the 0, 12, 24 weeks. The blood will be taken from the participant to test on biomarkers of cardio-metabolic risk which include Fasting insulin level, fasting glucose, triglyceride, cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No